CLINICAL TRIAL: NCT03735615
Title: Sprint Interval Training in Patients With Chronic Obstructive Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/723
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Exercise therapy; High-Intensity Interval Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: 10 patients with stable chronic obstructive lung disease (COPD) stage 3 and 4 according to GOLD guidelines (www.goldcopd.org), recruited from outpatient ward of the Lung Department at St Olav University Hospital. Control group of 10 age-matched but otherwise healthy subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chronic obstructive lung disease (Experimental)
  Interventions: Behavioral: sprint interval training
- healthy control (Experimental)
  Interventions: Behavioral: sprint interval training

INTERVENTIONS:
Behavioral: sprint interval training — Each training session will be performed 3 times per week for 3 weeks. Each session consists of 3-5x20 sec all-out cycling efforts against a load corresponding to 0.05-0.07 kg/kg body mass, separated by 3-5 min of low intensity cycling (20-50 W), on a lode bicycle ergometer (Excalibur Sport V2.0, Groningen, the Netherlands). All training sessions includes a 5 min warm-up and 3 min cool-down.

SUMMARY:
Exercise therapy is a cornerstone in the management of patients with Chronic Obstructive Pulmonary disease (COPD), and supervised walking exercise three times a week over 12 weeks improves walking ability and quality of life. Despite this, very few patients exercise on a regular basis. The underuse of exercise in COPD patients can partly be explained by discomfort during exercise because it evokes dyspnea, and thereby explain lack of participation in exercise. If the goal is to offer the best medical therapy to these patients, new and effective exercise training methods must be explored and defined since exercise training is an important part of pulmonary rehabilitation.

Intention is to study a new training method called sprint interval training (SIT), which consists of high intensity bouts with very short duration. The idea behind SIT is to avoid the dyspnea associated with traditional endurance training, thus maximizing exercise power without excessive discomfort. The investigators will study training adaptations in patients with COPD and compare the results with age-matched controls.

It is expected that both COPD-patients and healthy elderly will improve exercise cycle time until exhaustion after SIT training, and also that the improvement will be larger in the healthy group due to higher absolute training intensity.

ELIGIBILITY:
Inclusion Criteria (patients):

* stable CPOD stage 3 and 4 according to GOLD guidelines (www.goldcopd.org)
* post bronchodilator FEV < 50%

Exclusion Criteria:

* having participated in a pulmonary rehabilitation program during the last 3 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
exercise cycle time to exhaustion | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No